CLINICAL TRIAL: NCT06318000
Title: Assessment of the Relationship Between the Visual Impairment Degree and the Level of Children's Fundamental Motor Skills, Balance and Bilateral Coordination
Brief Title: Physical Activity and Sports for People With Visual Impairments
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: SN4/20/22
Record Dates: First submitted 2024-03-01; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Blindness; Visual Impairment
Keywords: Balance; Fundamental Motor Skills; Bilateral Coordination; Visual Impairments
MeSH Terms: conditions — Blindness; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons with visual impairments: Youth aged 7-17 years, male and female, with congenital or acquired visual impairment
  Interventions: Other: Balance test, bilateral coordination test, fundamental motor skills test
- Able bodied persons: Youth aged 7-17 years, male and female, without impairments
  Interventions: Other: Balance test, bilateral coordination test, fundamental motor skills test

INTERVENTIONS:
Other: Balance test, bilateral coordination test, fundamental motor skills test — Functional assessment

SUMMARY:
Purpose of this study was to assess the relationship between the visual impairment degree and the level of children's fundamental motor skills, balance and bilateral coordination.

DETAILED DESCRIPTION:
The participants were presented with the procedure of the study and informed that they could resign from their participation in the study at any stage. All participants legal guardians, were given the written informed consent form after the detailed written explanation of the risk and benefits resulting from participation in this study. Static balance was assessed using the portable AccuSway-Optimized (ACS-O) by AMTI stabilographic platform (ACS Model). The study participants performed the both feet 30 second, single 10 second left and right-leg stance with eyes open (EO), and both feet 30 second, left and right-leg stance with eyes closed (EC). If the first attempt was not successful, study participants were able to do the second attempt. The tests were conducted approximately 2 hours after a meal, in a sports outfit, in a specially designated room.

The functional assessment of locomotor skills will utilize the "locomotion" subtest, which is part of the Test of Gross Motor Development, Second Edition (TGMD-3) battery. In the selected "locomotion" subtest, the following movement tasks (locomotor skills) are assessed: Run, Gallop, Hop, Horizontal Jump, Skip, Slide.

The subtest 4 "Bilateral Coordination" of the Bruininks-Oseretsky Test of Motor Proficiency (BOT-2) was used in this study. The BOT-2 is an individually administered test that includes goal-directed activities to measure a wide range of motor skills in individuals aged 4 to 21 years. Participants performed seven items:

1. Touching Nose with Index Fingers - Eyes Closed
2. Jumping Jacks
3. Jumping in Place - Same Sides Synchronized
4. Jumping in Place - Opposite Sides
5. Pivoting Thumbs and Index Fingers
6. Tapping Feet and Fingers - Same Sides Synchronized
7. Tapping Feet and Fingers - Opposite Sides

ELIGIBILITY:
Inclusion Criteria:

* written consent form,
* visual impairment (diagnosed)
* intellectual norm.

Exclusion Criteria:

* nervous system disorders,
* structural changes within the musculoskeletal system
* and intellectual limitations.

Ages: 7 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Participants were 51 individuals with congenital or acguired visual impairments (26 girls and 25 boys) aged 7 to 17. The group of able-bodied peers consisted of 25 individuals (13 girls and 12 boys).
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Center of pressure (CoP) path length was measured | Baseline
  CoP displacement analysis is used to assess postural sway, based on which the balance control function can be assessed
Surface area of stabilogram was measured | Baseline
  Based on the analysis of the surface area of the stabilogram, the level of balance control can be assessed
Raw and scale score for each item | Baseline
  Based on this information, the level of bilateral coordination can be assessed. The assessment consists of 12 elements, with 6 aimed at assessing locomotion skills and the remaining 6 at object control skills. The locomotion component includes running, galloping, hopping, skipping, jumping, and sliding. The object control component includes striking stationary ball, stationary dribbling, catching, kicking, striking moving ball, and rolling ball. Each task is performed twice, with 1 point awarded for correct execution and 0 points for incorrect execution in every task's criteria. The total score from both trials indicates the final score for each task.
Qualitative performance criteria (points) | Baseline
  Based on this information, the level of fundamental motor skills level can be assessed. Raw score for each item was converted into point score rated on a scale of 0 to 3 or 4 points, in accordance to the study protocol, and the standardization of the test described in the manual of the BOT-2. The sum of raw scores from all the 7 items ranged from 0 to 24 points. The scale score was used to describe the examinee's level of proficiency on the subtest 4. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Body mass in kg | Baseline
  body mass
Body height in cm | Baseline
  height

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Morgulec - Adamowicz, Prof, Study Director — Józef Piłsudski University of Physical Education in Warsaw
Locations (1):
- University of Physical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Role of vision in static balance in persons with and without visual impairments — https://pubmed.ncbi.nlm.nih.gov/33541039/
- See also: Description Effects of sport on static balance in athletes with visual impairments — https://pubmed.ncbi.nlm.nih.gov/30421870/
- See also: Test of Motor Proficiency Second Edition (BOT-2): Compatibility of the Complete and Short Form and Its Usefulness for Middle-Age School Children — https://pubmed.ncbi.nlm.nih.gov/31065548/
- See also: Test of Gross Motor Development - 3 — https://sites.google.com/view/tgmd-3/home